CLINICAL TRIAL: NCT04354454
Title: Step Into Support for Endurance and Strength (SISTERS)
Acronym: SISTERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Alexi A. Wright, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-065
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Gynecologic Cancer
Keywords: Gynecologic Cancer; Mobile Health; Fitness Tracker; Survivorship; Quality of Life; Physical Activity; Feasibility Study; Pilot
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitbit (Active Comparator): After the screening procedures confirm participation in the research study. Participants randomized into Fitbit only group.
  -- Participants will track their daily steps for 4.5 months with use of a Fitbit
  The study interventions involved in this research are:
  * Fitbit (also known as a wearable accelerometer or fitness tracker)
  * Way to Health platform
  * Surveys/Interviews
  Interventions: Other: Fitbit
- Fitbit + Game + Support from a Teammate (Experimental): After the screening procedures confirm participation in the research study. Participants randomized into Fitbit + Game + Support from a Teammate.
  * Participants will select a step goal, use a Fitbit to track daily activity, and select a teammate (e.g. family member or friend) who they think will help them achieve their goals.
  * Participants will participate a 3-month game designed to increase activity and then followed for another 1.5 months to see if their increased activity can be maintained without the game.
  The study interventions involved in this research are:
  * Fitbit (also known as a wearable accelerometer or fitness tracker)
  * Help from a Teammate (i.e. friend or family member chosen to help reach goals, if applicable
  * Way to Health Platform
  * Surveys/Interviews
  Interventions: Other: Fitbit + Game + Support from a Teammate

INTERVENTIONS:
Other: Fitbit — Participants will select a daily step goal and track their steps every day for 4.5 months.
  Arms: Fitbit
Other: Fitbit + Game + Support from a Teammate — Daily Fitbit tracking for 4.5 months, divided into 2 parts.
  * 3 months on "active intervention" with Fitbit, a Game, and Support from a self-selected Teammate and pre-designed game.
  * 1.5 month follow-up period with Fitbit and social support teammate only
  Arms: Fitbit + Game + Support from a Teammate

SUMMARY:
The Step into Support for Endurance and Strength (SISTERS) research study is evaluating whether a mobile health game designed to increase physical activity is feasible and acceptable in patients with gynecologic cancers.

-SISTERS is testing a mobile health intervention can help increase physical activity. Participants will be randomized to receive either 1) a Fitbit or 2) a Fitbit + a game + help from a friend or family member whom you chose will help the participant reach their goals. (i.e. a Teammate).

DETAILED DESCRIPTION:
This study is a two-arm randomized controlled pilot study designed to test the feasibility and acceptability of using a wearable accelerometer (Fitbit) vs. a wearable accelerometer (FItbit) + a game designed to help participants increase physical activity + social support improves participants' average daily step counts.

Eligible Participants will be randomly assigned into 1 of 2 groups

1. Fitbit (wearable accelerometer) or
2. Fitbit (wearable accelerometer) + game + help from a self-selected teammate

The study interventions involved in this research are:

* Surveys/Interviews
* Fitbits (also known as a wearable accelerometers or fitness trackers)
* Way to Health Platform
* Help from a Teammate (i.e. a friend or family member that participants choose to help them reach their goals)

It is expected that about 50 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with a gynecologic cancer (ovarian, fallopian tube, primary peritoneal carcinoma, uterine, or cervical) who have completed cancer treatment ≥ 6 weeks prior.
* Own a smartphone (Android or iOS).
* Can read and provide informed consent in English.
* Do not have cognitive, visual, or orthopedic impairments that preclude participation, as evaluated by the research staff or oncology provider.
* Insufficiently active, as indicated by a score of <14 on the Leisure Score Index of Godin Leisure-Time Exercise Questionnaire (LSI).
* No future chemotherapy planned (except maintenance treatments; e.g. PARP inhibitors or endocrine therapy)

Exclusion Criteria:

* Patients already participating in a mobile health intervention.
* Patients who do not own a smartphone or computer to transmit data from the wearable tracker.
* Self-reported inability to walk 2 blocks (at any pace).
* Patients who are unable to identify a social support partner (i.e. family member, friend, or partner) to participate in the study (if selected for the intervention arm).
* The following special populations will be excluded from this research:

  * Adults unable to consent
  * Individuals who are not yet adults (infants, children, teenagers)
  * Pregnant women
  * Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Rate of Enrollment | 3 months
  Feasibility will be demonstrated if ≥50% eligible participants enroll
Rate of Completion | 3 months
  Feasibility will be demonstrated if ≥75% of eligible participants complete the post-baseline outcome assessments.
Burden Rate | 3 months
  Acceptability will be defined as: ≤20% of participants reporting high study burden and ≤10% study withdrawal.
Rate of Activity | 3 months
  Perceived effectiveness will be defined as ≥70% of participants indicate that study participation motivated them to increase their activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Alexi A Wright, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Northern Light Cancer Care, Brewer, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lifespan Comprehensive Cancer Center, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu